CLINICAL TRIAL: NCT01318434
Title: A Double-Blind, Paroxetine- and Placebo-Controlled Study of 50 mg/Day and 100 mg/Day of EB-1010 Among Outpatients With Major Depressive Disorder Who Have Responded Inadequately to Prior Selective Serotonin Reuptake Inhibitors (SSRIs) and Serotonin Norepinephrine Reuptake Inhibitors (SNRIs) (Triple Reuptake Inhibitor Anti-Depressant Effects - TRIADE Study)
Brief Title: A Paroxetine- and Placebo-Controlled Study of 50 mg/Day and 100 mg/Day of EB-1010 Among Outpatients With Major Depressive Disorder Who Have Responded Inadequately to Prior Selective Serotonin Reuptake Inhibitors (SSRIs) and Serotonin Norepinephrine Reuptake Inhibitors (SNRIs)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Euthymics BioScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EB-1010-301
Record Dates: First submitted 2011-03-09; First posted 2011-03-18 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-11

CONDITIONS: Major Depressive Disorder
Keywords: Outpatient
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 1-(3,4-dichlorophenyl)-3-azabicyclo-(3.1.0)hexane hydrochloride; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- EB-1010 25 mg BID (Experimental): Experimental Active
  Interventions: Drug: EB-1010 25mg BID
- EB-1010 50 mg BID (Experimental): Experimental Active
  Interventions: Drug: EB-1010 50mg BID
- SSRI/SNRI (Active Comparator): Active Comparator
  Interventions: Drug: SSRI Active
- EB-1010 0 mg BID (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EB-1010 25mg BID — capsule once daily
  Arms: EB-1010 25 mg BID
Drug: SSRI Active — Active Comparator
  Arms: SSRI/SNRI
Drug: EB-1010 50mg BID — Experimental Active
  Arms: EB-1010 50 mg BID
Drug: Placebo — Placebo comparator
  Arms: EB-1010 0 mg BID

SUMMARY:
The main research hypothesis for this study is that, among patients with Major Depressive Disorder (MDD) who have responded inadequately to treatment with SSRIs or SNRIs, the degree of improvement, as measured by the change from baseline of the Montgomery-Asberg Depression Rating Scale (MADRS)will be significantly greater among patients treated with EB-1010 (at the dose of 50 mg/day or 100 mg/day) than among those treated with placebo using the sequential parallel comparison design. The secondary research hypothesis for this study is that, among patients with MDD who have responded inadequately to treatment with SSRIs or SNRIs, the degree of improvement in depressive symptoms, as assessed by the MGH Cognitive and Physical Functioning Questionnaire (MGH CPFQ) will be significantly greater among those treated with EB-1010 (50 mg/day or 100 mg/day) than those treated with the SSRI paroxetine.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to give informed consent, (as required by IRB/IEC), prior to the initiation of any protocol required procedures.
* Patients must be able to understand the nature of the study, agree to comply with the prescribed dosage regimens, report for regularly scheduled office visits, and communicate to study personnel about adverse events and concomitant medication use.
* Patients with a diagnosis of major depressive episode as defined by DSM-IV-TR criteria, based on the SCID-CT29; their major depressive episode must be deemed "valid" using the SAFER criteria interview24 administered by remote, independent raters.
* Patients who have reported a history for the current depressive episode of an inadequate response to 1 and no more than 1 adequate SSRI or SNRI treatment. An inadequate response is defined as less than a 50% reduction in depressive symptom severity, as assessed by the MGH ATRQ administered by remote, independent raters. An adequate trial is defined as an antidepressant treatment for at least 8 weeks duration at least at the minimum dose as specified in the MGH ATRQ.
* Patients must have a 17-item Hamilton Rating Scale for Depression (HAM-D-17) (whose score is derived from the HAM-D-28)20 score ≥ 18 during the screening phase to qualify for inclusion. The HAM-D-28 will be administered by the study clinicians at the screening and baseline visits, and by remote, independent raters during the screening phase at the time of the SAFER interview.
* Patients must have a Body Mass Index (BMI) of approximately 18-40.
* Patients must be able to be reliably rated on the psychiatric scales required by the protocol based on Investigator's judgment.
* Patients must be able to understand and read English.
* Placebo non-responders are defined as those patients who failed to achieve at least a 50% decrease in their MADRS score at visit 8 (Week 6), AND have a MADRS score of = or > 16 at visit 8 (Week 6)
* Men and women, ages 18 to 65 inclusive.
* Meet DSM-IV-TR criteria (by Structured Clinical Interview for DSM-IV-TR - SCID-CT) for MDD, current.
* Treated with one of the allowed SSRIs or SNRIs at adequate doses (defined as 20mg/day or more of citalopram; 10 mg/day or more of escitalopram, 50mg/day or more of sertraline; 125 mg/day or more of venlafaxine; 60 mg/day or more of duloxetine) during the current episode for at least 8 weeks, with the same, adequate dose over the last 4 weeks.
* Between the screen and baseline visits, patients must be documented to have less than a 25% reduction in QIDS-SR score.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of investigational product in such a manner that the risk of pregnancy is minimized. Adequate methods are defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectable or patch hormonal contraception, oral contraceptives, an IUD, double-barrier contraception, sexual abstinence. Form of birth control will be documented at screening and baseline.

WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea ³ 12 consecutive months); or women on hormone replacement therapy [HRT] with documented serum follicle stimulating hormone [FSH] level > 35 mIU/mL). Even women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential. WOCBP must have a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of investigational product.

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period [and for up to 4 weeks after the last dose of investigational product.
* WOCBP using a prohibited contraceptive method that does not meet established and acceptable medical standards.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to investigational product administration.
* Sexually active fertile men not using effective birth control if their partners are WOCBP.
* Patients who do not report any prior inadequate response (equal or greater than 50% decrease in depressive symptom severity) or report an inadequate response (less than 50% decrease in depressive symptom severity) to more than 1 prior adequate trials of antidepressant treatments during the current depressive episode (including monotherapy treatment and distinct combination regimens) at a therapeutic dose (as defined by the MGH ATRQ)22-23 and for an adequate duration (minimum 6 weeks for any monotherapy).
* Patients who report treatment with adjunctive medication (buspirone, atypical antipsychotics, lithium) to their antidepressant therapy for a minimum of 4 weeks during the current depressive episode.
* Patients with a current need for involuntary commitment or who have been hospitalized within 4 weeks of the Screening Visit for the current major depressive episode.
* Subjects with other DSM-IV-TR Axis I disorders other than Generalized Anxiety Disorder (GAD: 300.02), Social Anxiety Disorder (300.23), or Specific Phobia (300.29). Subjects with co-morbid GAD, Social Anxiety Disorder, or Specific Phobia are ineligible if the co-morbid condition is clinically unstable, requires treatment, or has been the primary focus of treatment within the 6 month period prior to screening. More specifically, patients who have a current Axis I diagnosis
* Patients experiencing hallucinations, delusions, or any psychotic symptomatology in the current or any previous depressive episode.
* Patients who have met DSM-IV-TR criteria for any significant substance use disorder within the past six months, based on the SCID-CT.
* Patients receiving new-onset psychotherapy and/or somatic therapy (light therapy, trans-cranial magnetic stimulation) within 6 weeks of screening, or at any time during participation in the trial.
* Patients who, in the opinion of the Investigator, are actively suicidal and at significant risk for suicide.
* Patients who have participated in any clinical trial with an investigational drug or device within the past month.
* Patients who routinely perform shift work and whose sleep-wake cycle is frequently changed because of their work.
* Patients who have received ECT in the past 20 years or Vagal Nerve/Deep Brain Stimulation during their lifetime.
* Unstable medical illness including, cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease.
* Subjects with evidence or history of significant neurological disorder, including head trauma with loss of consciousness, history of stroke, Parkinson's disease, epilepsy disorder, conditions that lower seizure threshold, seizures of any etiology (including substance or drug withdrawal), who are taking medications to control seizures, or who have increased risk of seizures as evidenced by history of EEG with epileptiform activity (with the exception of juvenile febrile seizures).
* Subjects who are known to have AIDS or to be HIV positive.
* Patients with a significant history of drug or food allergy or hypersensitivity. Specifically, patients who report a history of drug-induced and/or food-induced asthma, facial-swelling, tongue swelling, angioedema, urticaria, stridor, hives, epiglottis swelling, recurrent skin rashes, toxic epidermal necrolysis, or Stevens-Johnson Syndrome.
* Patients who, in the Investigator's judgment represent a significant risk of committing suicide during the course of the trial based on history or evaluation of current mental status. Patients with significant hostility and history of aggressive acts who, in the Investigator's judgment, represent a significant risk of committing violent acts during the course of the trial based on history or evaluation of current mental status.
* Patients who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the course of the trial.
* Patients with thyroid pathology (unless condition has been stabilized with medications for at least the past three months).
* Patients with a lifetime history of serotonin syndrome.
* Patients with a significant history of a seizure disorder.
* Patients who have received a vaccination in the past three months.
* Patients with a recent (within two weeks) viral or systemic illness.
* Patients with current skin rashes.
* Patients who have recently (within two weeks) begun any medications.
* Patients who have a positive urine drug screen which cannot be explained by prescribed medications.
* Patients with AST and/or ALT >2x ULN at the screening visit.
* Patients with abnormal thyroid-stimulating hormone (TSH) concentrations or positive hepatitis tests.
* Patients with clinically significant laboratory abnormalities (hematology, chemistry, urinalysis) or with Safety Values of Potential Clinical Concern (see Table 3).
* Diastolic blood pressure > 105 mmHg at screen or baseline.
* Any signs or symptoms that are, in the Investigator's judgment, medically significant, in that they would impact the patient's safety.
* Patients with a QTc value of 460 ms or greater.
* Patients who are known to be allergic or hypersensitive to paroxetine and EB-1010.
* Patients previously treated with and not responding to paroxetine
* Monoamine oxidase inhibitors (e.g., Nardil, phenelzine, Parnate, tranylcypromine, Marplan, isocarboxazide) treatment within the 2 weeks prior to enrollment.
* Patients who would likely require prohibited concomitant medications and/or other depression treatment during the trial.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.
* Patients who demonstrate a 25% or greater decrease in depressive symptoms as reflected by the QIDS-SR19 total score from screen visit to baseline visit.
* Patients who plan to have elective surgeries during the course of the study.
* Patients with a history of antidepressant-induced hypomania or dysphoria.
* Patients who demonstrate a less than 80% compliance (as measured by pill count) of their antidepressant medication during the Screening Phase.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in MADRS Score | 6 weeks
  Improvement in MADRS Score

SECONDARY OUTCOMES:
Change in Clinical Global Severity Scale | 6 weeks
  Degree of clinical global severity improvement

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tran, MD, Study Director — Euthymics BioScience, Inc.
Locations (43):
- United States (43):
  - Pacific Clinical Research Medical Group, Arcadia, California
  - Southwest Research, Inc., Beverly Hills, California
  - Synergy Clinical Research Center, National City, California
  - Clinical Innovations, Inc., Santa Ana, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Radiant Research, Inc., Denver, Colorado
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Sanitas Research, Coral Gables, Florida
  - Clinical Neuroscience Solution, Inc., Jacksonville, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Medical Research Group of Central Florida, Sanford, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - AMR Baber Research, Naperville, Illinois
  - Psychiatric Medicine Associates, Stokie, Illinois
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Clinical Insights, Glen Burnie, Maryland
  - Cambridge Health Alliance, Cambridge, Massachusetts
  - AccelRx Research, Fall River, Massachusetts
  - St Charles Psychiatric Associates, Saint Charles, Missouri
  - Global Medical Institutes, Princeton, New Jersey
  - CRI Worldwide, LLC, Willingboro, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - Community Research, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - North Star Medical Research, Middleburg Heights, Ohio
  - Neurology and Neuroscience Center of Ohio, Toledo, Ohio
  - SP Research, PLLC, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Southeastern PA Medical Institute, Broomall, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Scranton Counseling Center, Scranton, Pennsylvania
  - Radiant Research, Greer, South Carolina
  - Clinical NeuroScience Solutions, Inc., Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Radiant Research, Inc., Murray, Utah
  - Aspen Clinical Research, Orem, Utah
  - VCU, Richmond, Virginia
  - Dean Foundation for Health, Research & Education, Middleton, Wisconsin